CLINICAL TRIAL: NCT07395531
Title: Effect of Repetitive Bihemispheric Anodal Transcranial Direct Current Stimulation on Motor Function of Patients With Parkinson's Disease
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Ram Manohar Lohia Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Ashish Kumar Duggal, Professor, Department of Neurology, ABVIMS and Dr RML Hospital, New Delhi, Dr. Ram Manohar Lohia Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IEC/ABVIMS/RMLH/1092
Record Dates: First submitted 2026-01-25; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: PARKINSON DISEASE (Disorder); Parkinson Disease
Keywords: tDCS; Parkinson's Disease; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS arm (will receive true tDCS) (Experimental): Will receive true anodal tDCS stimulation
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS arm (will receive Sham stimulation) (Sham Comparator): Will not receive anodal tDCS stimulation
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Anodal tDCS stimulation
  Other Names: tDCS
  Arms: Anodal tDCS arm (will receive true tDCS)
Device: Transcranial Direct Current Stimulation — Sham tDCS
  Other Names: tDCS
  Arms: Sham tDCS arm (will receive Sham stimulation)

SUMMARY:
Dopaminergic medications and Deep Brain Stimulation (DBS) are the current standards interventions for Parkinson's Disease. Pharmacotherapy with dopaminergic drugs leads to partial improvement in motor functions of patients. Invasive therapies like DBS have as yet limited availability and accessibility, with risk of adverse events as well. Non invasive therapies like Transcranial Direct Current Stimulation (tDCS) are currently increasingly being probed for their therapeutic value, in view of their safety, portability and convenience of administration.

Improvement in motor function immediately after a single session of tDCS has been observed. The effect of single simulation is not sustained beyond a few days. Only few studies with varied sites of stimulation have evaluated the effect of repetitive tDCS on motor function improvement in patients with Parkinson's Disease, with conflicting results. There is an unmet need to probe the utility of repetitive tDCS on motor function of patients with Parkinson's Disease.

We aim to probe the effect of repetitive tDCS of dorsolateral prefrontal cortex and M1 cortex on motor function in patients with Parkinson's Disease (Hoehn and Yahr stage 2 to 4).

ELIGIBILITY:
Inclusion Criteria:

1. Patients fulfilling the Movement Disorder Society (MDS) clinical diagnostic criteria for Parkinson's disease.
2. Patients with Hoehn & Yahr stages 2-4 Parkinson's disease.
3. Patients maintained on stable medical regimen for at least 1 month before entering the study.

Exclusion Criteria:

1. Patients with other confounding neurological and psychiatric disorders.
2. The presence of metal objects or stimulators in the head.
3. Patients with a history of deep brain stimulation.
4. Patients with history of seizures.
5. Patients with skull defect due to surgery e.g. craniectomy
6. Patients with scalp condition likely to obstruct application of electrodes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
To determine change in motor function score as assessed by Movement Disorder Society - Unified Parkinson's Disease Rating Scale Part - III scale 1 week after the repetitive tDCS (Minimum Score 0, Maximum Score 132, higher scores indicate more disability) | 1 week

SECONDARY OUTCOMES:
To determine the change in Timed Up and Go test score of patients with Parkinson's Disease at 1 week after the repetitive tDCS (higher times indicate disability with increased risk of fall) | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Kumar Duggal, DM (Neurology), Principal Investigator — Atal Bihari Vajpayee Institute of Medical Sciences and Dr. Ram Manohar Lohia Hospital, New Delhi
Locations (1):
- Atal Bihari Vajpayee Institute of Medical Sciences and Dr. Ram Manohar Lohia Hospital, New Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
IPD collected throughout the trial will be available from the Principle Investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF

DOCUMENTS (4):
  • Study Protocol: Study Protocol Version with corrections (2026-01-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT07395531/Prot_000.pdf
  • Study Protocol: Study Protocol Original (2026-01-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT07395531/Prot_001.pdf
  • Informed Consent Form: Informed Consent with Corrections (2026-01-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT07395531/ICF_002.pdf
  • Informed Consent Form: Informed Consent Original (2026-01-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT07395531/ICF_003.pdf